CLINICAL TRIAL: NCT06485531
Title: The Effect of Pranayama and Pursed Lip Breathing Exercise on Pain and Respiration After Coronary Bypass Surgery
Brief Title: The Effect of Pranayama on Pain and Respiration After Coronary Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tugba ALBAYRAM, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: TALBAYRAM
Record Dates: First submitted 2024-06-18; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Respiratory; Postoperative Pain; Nursing
Keywords: CABG, pranayama, pain, respiration, nursing
MeSH Terms: conditions — Pain, Postoperative; Pain; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pranayama (Active Comparator): Nadi Shothana Pranayama was applied to the patients for 15 minutes before the surgery and for 7 days after the surgery. After the application, FVC, FEV1, and FEV1/FVC values were measured with a spirometer (Contec Spirometer SP70B, Contec Medical Systems Co,. Ltd., China) and recorded in the Patient Follow-up Form. In cases where the patient did not perform well, the measurement was repeated at least three times and the best data was taken. Systolic and diastolic blood pressure, heart rate, respiratory rate, and peripheral oxygen saturation, which were thought to affect the results of FVC, FEV1, and FEV1/FVC values, were also measured and recorded. In addition, hematocrit level, analgesia dose, and amounts used during the day were recorded daily and in the Patient Follow-up Form. Pain levels were evaluated 4 times daily (10:00-14:00-22:00-06:00) during the 0th to 6th days after surgery and recorded on the Visual Analog Scale Form.
  Interventions: Other: Pranamaya
- Pursed Lips Breathing (Sham Comparator): Pursed Lip Breathing Exercise was applied to the patients before and after the surgery for 15 minutes. After the application, FVC, FEV1, and FEV1/FVC values were measured with a spirometer (Contec Spirometer SP70B, Contec Medical Systems Co., Ltd., China) and recorded in the Patient Follow-up Form. (Annex-3). In cases where the patient did not perform well, the measurement was repeated at least three times and the best data was taken. Systolic and diastolic blood pressure, heart rate, respiratory rate, and peripheral oxygen saturation, which are thought to affect the results of FVC, FEV1, and FEV1/FVC values, were also measured and recorded before and after the application. In addition, hematocrit level, analgesia dose, and amounts used during the day were recorded daily and in the Patient Follow-up Form. Pain levels were evaluated 4 times daily (10:00-14:00-22:00-06:00) during the 0th to 6th days after surgery and recorded on the Visual Analog Scale Form.
  Interventions: Other: Pursed Lips Breathing
- Control (No Intervention): No intervention was made to the control group patients. FVC, FEV1 and FEV1/FVC values of the patients were measured with a spirometer (Contec Spirometer SP70B, Contec Medical Systems Co., Ltd., China) before the surgery and for 7 days after the surgery. In cases where the patient did not perform well, the measurement was repeated at least three times and the best data was taken. Systolic and diastolic blood pressure, heart rate, respiratory rate, and peripheral oxygen saturation, which are thought to affect the results of FVC, FEV1, and FEV1/FVC values, were also measured and recorded at 15-minute intervals. In addition, the hematocrit level, the dose, and amount of analgesia used during the day were recorded daily and in the Patient Follow-up Form. Pain levels were evaluated 4 times daily (10:00-14:00-22:00-06:00) during the 0th to 6th days after surgery and recorded on the Visual Analog Scale Form.

INTERVENTIONS:
Other: Pranamaya — Pranamaya
  Arms: Pranayama
Other: Pursed Lips Breathing — Pursed Lips Breathing
  Arms: Pursed Lips Breathing

SUMMARY:
After CABG surgery, patients tend to breathe superficially because they experience pain while breathing. By restricting deep inspiration and cough; There is a decrease in lung tidal volume, vital capacity, and functional residual capacity. Accordingly, alveolar ventilation also decreases, and the oxygenation levels of the organs decrease due to alveolar collapse or developing hypoxemia. Due to the pain experienced, patients cannot cough and secretions accumulate in the alveoli. Due to accumulated secretions, patients are more prone to atelectasis and lung infections. The risk of pulmonary embolism increases in patients due to the limitation of movement caused by pain. It is aimed to replace these weak breathing patterns with conscious breathing patterns provided by pranayama. While pranayama improves regular, slow, and deep breathing, it activates nasal breathing and provides diaphragmatic breathing. Thanks to the suction pressure created in the chest cavity with diaphragmatic breathing, the venous return of blood also improves. Along with all these changes, it also helps reduce the heart's workload by regulating circulatory functions such as blood pressure, heart rate, left ventricular pressure, and coronary artery diameter. Alternating nasal breathing, slow and deep breathing, applied during pranayama, helps relieve breathing work in eliminating excessive breathing patterns. In addition, nasal breathing balances sympathetic and parasympathetic activity and makes an important contribution to the regulation of the activities of the autonomic nervous system. The vagus nerve, which has a parasympathetic effect, stimulates the left nostril, diagram, stomach, hypothalamus, pineal gland, and suprachiasmatic nucleus and stimulates the diaphragm and stomach, and with this control of the autonomic nervous system, it helps to keep the respiratory rate within normal ranges, improve breathing, reduce stress hormones and help relaxation. Controlled inspiration, breath holding, and slow expiration practices performed with pranayama also contribute to increasing the general capacity of the lungs and gradually improving respiratory functions.

ELIGIBILITY:
Inclusion Criteria:

* CABG surgery performed on a stopped heart (On pump),
* Cardiopulmonary risk index score ≤2
* Those aged 18 and over,
* Being literate and communicative,
* American Society of Anesthesiologists (ASA) classification I or II,
* Preoperative respiratory function tests with normal FEV1, FVC, FEV1/FVC values,
* No complications developed during and after the surgical intervention,
* An analgesic drug with the same active ingredient is applied to control pain after surgical intervention,
* Patients who were administered antibiotics with the same active ingredient after surgical intervention were included.

Exclusion Criteria:

* CABG surgery performed on a working heart (off-pump),
* Cardiopulmonary risk index score ≥4
* Complications developing during or after surgery,
* Intubated,
* Those with chronic pain in the pre-surgical period,
* Those with limited movement activity before surgery,
* Having a body mass index (BMI≥30),
* Patients who could not adapt to and tolerate the pranayama technique were not included in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
postoperative FVC | From admission to discharge, up to 1 week
  Improvement in FVC in patients treated with Pranayama after CABG
FEV1 | From admission to discharge, up to 1 week
  Improvement in FEV1 in patients treated with Pranayama after CABG
FEV1/FVC level | From admission to discharge, up to 1 week
  Improvement in FEV1/FVC level in patients treated with Pranayama after CABG
Change in postoperative pain measured by VAS | From surgery to 3 days after surgery
  Change in postoperative pain measured by VAS in patients who underwent pranayama after CABG

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Albayram, Principal Investigator — University of Gaziantep
Locations (1):
- Tuğba Albayram, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be made available to other researchers